CLINICAL TRIAL: NCT00458185
Title: Multicentre, Open-Labeled Study Of Etanercept In The Treatment Of Patients With Ankylosing Spondylitis
Brief Title: Study Evaluating Etanercept in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0881A-101871
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: etanercept

SUMMARY:
This study will assess the efficacy of etanercept for the treatment of Ankylosing Spondylitis (AS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AS, as defined by Modified New York Criteria for Ankylosing Spondylitis, aged between 18 and 70 years of age.
* BASDAI greater than or equal to 40 (all scores on a scale of 0 to 100).
* Negative result of serum human chorionic gonadotropin (HCG) pregnancy test taken at screening in all women except those surgically sterile or at least 1 year postmenopausal.

Exclusion Criteria:

* Complete ankylosis (fusion) of spine.
* Previous receipt of etanercept, antibody to TNFα, or other TNFα inhibitors.
* Use of disease modifying antirheumatic drugs (DMARDs) other than hydroxychloroquine, sulphasalazine, and methotrexate within 4 weeks of baseline. Patients treated with hydroxychloroquine, sulphasalazine, and methotrexate may continue these drugs during this study but doses must be held stable for 4 weeks before baseline examination and for the duration of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-08; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of etanercept (25 mg, twice weekly) based on the percentage of patients who achieve the Assessment in Ankylosing Spondylitis (ASAS) Response Criteria at 20% level at week 12.

SECONDARY OUTCOMES:
Efficacy at 50% and 70% levels week 12; frequency and time to partial remission; safety; patient and physician global assessment, nocturnal and total back pain, BASFI, BASDAI; spinal mobility; complete joint assessment; hip involvement; ESR, CRP.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer